CLINICAL TRIAL: NCT06372808
Title: The Effect of Plyometric Exercises on Physical Fitness Parameters in Freestyle Adolescent Wrestlers
Brief Title: The Effect of Plyometric Training in Freestyle Adolescent Wrestlers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Talha gökçe, İnvestigator, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/118
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2023-12

CONDITIONS: Physical Fitness; Power
Keywords: Plyometric Exercises; Physical Fitness; Wrestlers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training Group (Experimental): The training group will receive a carefully designed plyometric training program by a qualified and experienced physiotherapist. This program will be implemented twice a week for eight weeks, with the number of sets and repetitions of the exercises adjusted weekly to ensure a progressive and safe training regimen. Evaluations will be conducted at the beginning and end of the eight weeks to assess the effects of the plyometric training.
  Plyometric training program:
  * Vertical jumps
  * Tuck jumps
  * Two-legged broad jumps
  * One-legged bounding
  * Depth jumps from a 40 cm height
  Rest intervals between repetitions and sets were set at 15-30 seconds. A 20-minute warm-up period before the program and a 20-minute cool-down period afterwards were planned.
  Interventions: Other: The Plyometric Exercise
- Control Group (Experimental): The control group will continue their regular training program without additional interventions. The routine training program for the control group includes basic strength training (weightlifting exercises), cardiovascular training (biking, running, sprint training, jogging), technical and tactical training, and match-style wrestling. Evaluations will be conducted at the beginning and end of the eight weeks.
  Interventions: Other: The Regular Training

INTERVENTIONS:
Other: The Plyometric Exercise — The training group will perform plyometric exercises for eight weeks in addition to their regular training program.
  Arms: Training Group
Other: The Regular Training — The control group's regular training includes basic strength training, cardiovascular training, technical and tactical training, and match-style wrestling.
  Arms: Control Group

SUMMARY:
This study aims to determine the effect of plyometric exercises on physical fitness parameters in freestyle adolescent wrestlers.

DETAILED DESCRIPTION:
Plyometric exercises are an effective training method that converts strength gains into power by applying specific power (explosive force) training. Plyometric training also dramatically contributes to converting acquired strength into wrestling-specific power. In light of this information, the relatively scarce literature on plyometric training with wrestlers, particularly adolescent freestyle wrestlers, will be studied. This study examines the effects of different plyometric training on physical fitness parameters in adolescent freestyle wrestlers over eight weeks.

The investigators will involve participants who meet the inclusion criteria and who will be randomly assigned to either the control or training group. The training group will undergo plyometric exercise training twice a week for eight weeks in addition to their regular training program. Conversely, the control group will continue their regular training program without additional interventions. Evaluations will be conducted at the beginning and end of the eight weeks to assess the effects of the plyometric training.

The routine training program for the control group participants includes basic strength training (weightlifting exercises), cardiovascular training (biking, running, sprint training, jogging), technical and tactical training, and match-style wrestling. The plyometric training program will be implemented twice a week for 8 weeks, with the number of sets and repetitions of the exercises adjusted weekly to ensure a progressive and safe training regimen.

The investigators will assess the evaluation criteria at the beginning and end of the 8-week training period, comparing pre- and post-training data and conducting intergroup comparisons. Two measurements will be recorded according to these parameters. By the end of the study, the investigators will provide a comprehensive analysis of the impact of the plyometric training program on the physical fitness parameters of freestyle adolescent wrestlers, supported by robust data.

ELIGIBILITY:
Inclusion criteria for the study:

* Individuals engaged in freestyle wrestling sport with a valid license,
* Aged between 10 and 15 years old,
* Have been practicing this sport for at least three years,
* Not involved in any other sports discipline,
* Willing to cooperate and volunteer for the study,
* The research will include those who have not received medical treatment in the last three months and will not receive treatment during the study period.

Exclusion criteria for the study:

* Individuals with injuries and chronic pain,
* Smokers,
* Regular medication users,
* Those with neurological and systemic diseases,
* Individuals who have experienced trauma and undergone surgery in the last three months,
* Athletes who withdraw their voluntary participation

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Strength at 8 weeks | Baseline, 8 weeks
  Hand Grip Strength Test: Grip strength is a measurement method to evaluate overall body strength and upper extremity performance. This test measures the maximum isometric contraction strength of the hand and forearm muscles. It will be conducted using a hand-grip dynamometer.
  Back and Leg Strength Test: This test assesses the strength of the back and leg muscles. It is performed using a back-leg dynamometer.
Change from Baseline in Endurance at 8 weeks | Baseline, 8 weeks
  The McGill Core Endurance Test, which consists of four positions (Trunk Flexors Endurance Test, Trunk Extensors Endurance Test, and Right and Left Lateral Plank Tests), will measure participants' endurance. The maximum time each participant can remain in these positions will be recorded in seconds.
  Collectively, these tests evaluate the endurance and strength of various core muscles.
Change from Baseline in Agility at 8 weeks | Baseline, 8 weeks
  Agility will be measured using the Agility T-Test. This test is set up in a T-shape with four contact points, covering a 10-meter length and width area. Participants must complete a series of movements between these contact points in different directions and patterns as quickly as possible. What sets this test apart from other agility tests is that the participant always faces the same direction. Changes in direction are made by sidestepping to the right and left or by running backward.
Change from Baseline in Wrestling Performance at 8 weeks | Baseline, 8 weeks
  Wrestling performance will be measured using a special judo fitness test. The test consists of three application sections of 15, 30, and 30 seconds each, with 10-second rest intervals between applications. In each section, the judoka (tori) must throw the other two judokas (uke) as quickly as possible using the ipon-seoi-nage technique. The distance between the ukes is 6 meters, and the tori starts the applications at 3 meters from each uke.
  Participants' heart rates (HR) are recorded immediately after the test (HR_post) and one minute later (HR_1 min). The throws and HR are recorded at the end of the test.
  The scoring index for this test is a combination of your post-test and 1-minute later heart rates, divided by the total number of throws. The formula is as follows: Index score = (HR_post + HR_1 min) / throws (total).

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Tuncer, PhD, Study Director — Hasan Kalyoncu University
Locations (1):
- Batipark Sports Hall, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No